CLINICAL TRIAL: NCT05305079
Title: Non-Arteritic Anterior Ischemic Optic Neuropathy Risk Factors: New Perspectives
Brief Title: NA-AION Risk Factors: New Perspectives
Acronym: NARROW
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Velux Fonden (Other); Fight for Sight (Other); University of Copenhagen (Other); Hamilton Health Sciences Corporation (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Farabi Eye Hospital (Other); Wellington Hospital (Other Government); University of Colorado, Denver (Other); University of Utah (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); University of Sydney (Other); Stanford University (Other); Moorfields Eye Hospital NHS Foundation Trust (Other); Massachusetts Eye and Ear Infirmary (Other); University Hospital, Bordeaux (Other); Synoptik-Fonden (Unknown)
Responsible Party: Principal Investigator, Steffen Hamann, MD, PhD, associate professor, Rigshospitalet, Denmark
Other Study IDs: H-20073063
Record Dates: First submitted 2021-07-26; First posted 2022-03-31 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2022-03

CONDITIONS: Non-arteritic Ischemic Optic Neuropathy; Optic Disk Drusen
Keywords: Optical Coherence Tomography; Optical Coherence Tomography Angiography
MeSH Terms: conditions — Optic Disk Drusen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ODD-AION: NA-AION patients with ODD aka. Optic disc drusen associated non-arteritic anterior ischemic optic neuropathy.
- nODD-AION: NA-AION patients without ODD aka Non-optic disc drusen associated non-arteritic anterior ischemic optic neuropathy.

SUMMARY:
The purpose of the study is to use new diagnostic methods (OCT and OCT-A) to shed light on risk factors for the development of NA-AION. The risk factors we are focusing on are comorbidities along with anatomical and vascular characteristics of the optic nerve.

DETAILED DESCRIPTION:
Non-arteritic anterior ischemic optic neuropathy (NA-AION) is the most common acute optic neuropathy in the middle-aged and elderly population and can also occur in children and young adults. NA-AION leads to irreversible vision loss, and there is currently no effective treatment. In recent years, acellular calcified deposits in the optic nerve head called optic disc drusen (ODD) have been investigated as an important risk factor for NA-AION in patients under the age of 50.

The purpose of the study is to use new diagnostic methods optical coherence tomography (OCT) and OCT-angiography (OCTA) to shed light on risk factors for the development of NA-AION. We will perform two sub-studies:

1. Characteristics of the optic nerve head anatomy including the presence of ODD as risk factors for the development of NA-AION.
2. Vascular comorbidities and in vivo vasculature as a risk factor for developing NA-AION.

The study is an international prospective multicenter study including 20 sites in 9 different countries. The study population is patients diagnosed with NA-AION in a 1.5-year inclusion period. Each included patient gets 1-2 follow up visits during a 3-month follow up time.

Included patients will be examined as per standard clinical care for that site including OCT and OCT-A. Standard clinical care includes at least: obtaining medical history, measurement of visual acuity, slit lamp examination, and automated perimetry.

Characteristics and risk factors in NA-AION patients with ODD (ODD-AION) will be compared with NA-AOIN patients without ODD (nODD-AION).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of first episode of NA-AION in study eye with symptom onset within 1 month prior
2. Subject age: Age >10
3. NA-AION diagnosis requires:

   * disc edema seen by site PI or by referring doctor
   * visual field defect in the study eye consistent with NA-AION and mean deviation worse than 3.0 dB using the study visual field examination protocol
   * relative afferent pupillary defect (unless the fellow eye had previous NA-AION or other optic nerve or retinal disease that is not exclusionary)

Exclusion Criteria:

1. Previous episode of NA-AION in the study eye only
2. Intraocular pressure of >21 mm Hg in the study eye
3. Clinical or pathological evidence of giant cell arteritis
4. Diseases that may affect the optic nerve: glaucoma, multiple sclerosis, Alzheimer disease, and Parkinson disease. Evidence of optic disc drusen and optic nerve hypoplasia are not exclusion criteria given they are important parts of the study. We will not exclude significant retinal diseases, since they may be related to underlying etiologies giving rise to ODD, such as macular degeneration, retinal dystrophies, but eyes with significant retinal diseases will be analyzed separately.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is patients diagnosed with NA-AION in a 1.5-year inclusion period.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Anatomical characteristics on OCT | At enrollment
  Presence of ODD. Diameter of the scleral canal, disc area and rim on each quadrant of the optic disc, thickness of the peripapillary choroid, presence of peripapillary hyperreflective ovoid mass-like structures, and prelaminar hyperreflective lines.
Anatomical characteristics on OCT | 3-months follow-up visit
  Presence of ODD. Diameter of the scleral canal, disc area and rim on each quadrant of the optic disc, thickness of the peripapillary choroid, presence of peripapillary hyperreflective ovoid mass-like structures, and prelaminar hyperreflective lines.
Vascular characteristics on OCT-A | 3-months follow-up visit
  Transient versus persistent findings of ischemia, segmental location and extent of reduced vessel density. If ODD is present the vessel density will be compared to ODD location and volume.

SECONDARY OUTCOMES:
ODD characteristics | At 3-months follow-up visit
  If ODD is present the volume and location of the ODD (superficial vs. deep) is measured using 3D-segmentation
Best corrected visual acuity | At enrollment
  Assessed on Snellen or ETDRS chart
Best corrected visual acuity | 3-months follow-up visit
  Assessed on Snellen or ETDRS chart
Visual field test | At enrollment
  Autoperimetry: SITA fast or standard 24-2
Visual field test | 3-months follow-up visit
  Autoperimetry: SITA fast or standard 24-2
Questionnaire score: NEI-VFQ-25 including 10-item NO supplement score | At enrollment
  Score on questionnaire: National Eye Institute Visual Function Questionnaire 25 and 10-item Neuro-Ophthalmic Supplement
  A vision-targeted composite score of the NEI-VFQ-25 together with the 10-item NO supplement score is calculated. The scale is 0-100 where a high score represents better functioning.
Questionnaire score: NEI-VFQ-25 including 10-item NO supplement score | 3-months follow-up visit
  Score on questionnaire: National Eye Institute Visual Function Questionnaire 25 and 10-item Neuro-Ophthalmic Supplement.
  A vision-targeted composite score of the NEI-VFQ-25 together with the 10-item NO supplement score is calculated. The scale is 0-100 where a high score represents better functioning.
Prevalence of comorbidities | At enrollment
  ischemic heart disease, stroke (ischemic or hemorrhagic), arterial hypertension, diabetes mellitus, end stage renal disease, smoking (now or previous), dyslipidemia, obstructive sleep apnea/continuous positive airway pressure (CPAP) use, phosphodiesterase-5 inhibitor use or ocular surgery.

OTHER OUTCOMES:
Eye refraction in diopters | At enrollment
  Spherical and cylindrical refraction. Measurements in diopters.
Color vision test score as fraction | At enrollment
  Assessed on Ishihara or Hardy-Rand-Rittler plates. Measured as the fraction of how many correct plates out how many plates are used in the assessment in total. A score of 0 means no plates were read correctly and 1 means all plates were read correctly.
Color vision test score as fraction | 3-months follow-up visit
  Assessed on Ishihara or Hardy-Rand-Rittler plates. Measured as the fraction of how many correct plates out how many plates are used in the assessment in total. A score of 0 means no plates were read correctly and 1 means all plates were read correctly.
Eye biometry: Axial length | At enrollment
  axial length of the eye in mm
Eye biometry: Keratometry | At enrollment
  The curvature of the cornea in diopters

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Hamann, Principal Investigator — Rigshospitalet, Denmark
Locations (20):
- United States (5):
  - Stanford Medicine, Palo Alto, California
  - UCSF Medical Center, San Francisco, California
  - University og Colorado, Boulder, Colorado
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - John A. Moran Eye Center, Salt Lake City, Utah
- Sydney Eye Hospital, Sydney, Australia
- Canada (3):
  - University of Calgary, Calgary
  - Research St. Joseph's, Hamilton
  - Lawson Health Research Institute, London
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
- Bordeaux University Hospital, Bordeaux, France
- Farabi Eye Hospital, Tehran, Iran
- Sheba Medical Center, Tel Aviv, Israel
- Capital and Coast DHB, Wellington, New Zealand
- United Kingdom (3):
  - University of Cambridge, Cambridge
  - King's College Hospital, London
  - Moorfield's Eye Hospital, London

REFERENCES:
- [Derived] Klefter ON, Hansen MS, Lykkebirk L, Subhi Y, Brittain JM, Jensen MR, Dohn UM, Fana V, Wiencke AK, Heegaard S, Terslev L, Hamann S. Combining Paracentral Acute Middle Maculopathy and Peripapillary Fluid as Biomarkers in Anterior Ischemic Optic Neuropathy. Am J Ophthalmol. 2025 Mar;271:329-336. doi: 10.1016/j.ajo.2024.12.001. Epub 2024 Dec 6. PMID 39645178